CLINICAL TRIAL: NCT06385171
Title: Assessing the Impact of Botulinum Toxin Type A on Facial Wrinkles: A Comprehensive Clinical Investigation
Status: Recruiting | Type: Observational
Sponsor: Global Aesthetics LLC (Other)
Responsible Party: Principal Investigator, Otis Reid Scroggins, Director, Principal Investigator, Clinical Aesthetician, Global Aesthetics LLC
Other Study IDs: FFA-BTX-1
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Wrinkle
Keywords: Facial Wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Group Assignment: Experimental: Botulinum Toxin Type A:
  Patients will receive their first treatment on Day 1 after screening, with baseline facial muscle assessment on Day 0. Touch-up treatments will be given every 3 weeks until the sixth month. At Week 3, primary efficacy assessment will be conducted by evaluating facial movement control. Longevity assessment will occur at Month 6, with additional evaluation of immune response. This cycle will repeat for the second dose after six months until one year, and the same cycle will repeat for the 2nd dose.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — The intervention involves the administration of Botulinum Toxin Type A, with dosages regulated according to FDA guidelines. Each injection site will receive a maximum of 4 units, adhering to the FDA's recommended dosage limits. Dosages administered will be tailored to each patient's needs and will be recorded in their individual patient information chart.
  Other Names: OnabotulinumtoxinA

SUMMARY:
A study conducting to see how well a treatment called Botulinum Toxin Type A works for reducing facial wrinkles. The study will help us understand if this treatment is safe and effective for making wrinkles on the face less noticeable.

DETAILED DESCRIPTION:
The primary purpose of this clinical trial is to evaluate the efficacy and safety of Botulinum Toxin Type A in the treatment of facial wrinkles among a diverse population, with a specific aim to bridge the gap between cosmetic injectables and varying financial statuses of potential patients. This study intends to determine the degree to which Botulinum Toxin Type A can reduce the appearance of facial wrinkles, identify the optimal dosage for significant cosmetic improvement with minimal side effects, and assess patient satisfaction with the outcomes. By conducting a rigorous, controlled, and open label methodology, this research aspires not only to provide comprehensive data supporting the use of Botulinum Toxin Type A as a safe and effective treatment for aesthetic improvement but also to make such treatments more accessible and affordable. This endeavor seeks to democratize cosmetic enhancements, ensuring that individuals across different economic backgrounds can benefit from advancements in cosmetic dermatology. Ultimately, the study aims to offer valuable insights into cost-effective practices without compromising treatment quality, thereby enhancing patient care practices and contributing significantly to the field of cosmetic dermatology.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders.
* Must be in good physical health.
* Age between 20 and 65 years.
* Presence of both static (unchanging) and moderate dynamic (movement-induced) wrinkles on the forehead or glabellar region.
* Must possess the willingness and ability to understand and provide informed consent, as well as effectively communicate with study personnel.

Exclusion Criteria:

* Pregnant or breastfeeding female.
* Age below 20 or above 65 years.
* History of neuromuscular disorders, such as myasthenia gravis.
* History of facial surgery or presence of scars in the treatment area that could potentially interfere with or confound the results of the study.
* Recent treatment history within the past 6 months in the forehead or glabellar region, including:
* Ablative laser procedures.
* Radiofrequency device treatments.
* Ultrasound device treatments.
* Medium to deep chemical peels.
* Temporary soft tissue augmentation.
* Semi-permanent soft tissue augmentation within the past 2 years.
* Permanent soft tissue augmentation.
* Planned cosmetic procedures within the next 6 months in the same region.
* Intended use of tretinoin or retinoic acid within the next 6 months.
* Presence of active infection in the treated area, excluding mild acne.
* Allergy to cow's milk protein or albumin.
* Use of aminoglycoside medications.
* Current use of anticoagulation therapy.
* History of bleeding disorders.
* Diagnosis of mental illness.
* Inability to comprehend the study protocol or provide informed consent.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population from which the groups or cohorts will be selected consists of individuals aged between 20 and 65 years, regardless of gender, who are seeking treatment for facial wrinkles. These individuals must be in good physical health and exhibit both static (unchanging) and moderate dynamic (movement-induced) wrinkles on the forehead or glabellar region. They should also possess the willingness and ability to understand and provide informed consent for participation in the study. This population may include individuals from various backgrounds and demographics who are interested in cosmetic dermatology procedures.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Change in facial wrinkles and Lines | Upto 2 years
  Visual Assessment: The Principal Investigator (PI) will visually assess the change in wrinkles and lines on the patient's face compared to baseline, using the following grading scale:
  Grade 0: No improvement in wrinkles. Grade 1: Minimal improvement, slight reduction in wrinkles. Grade 2: Moderate improvement, noticeable reduction in wrinkles. Grade 3: Significant improvement, substantial reduction in wrinkles.
  Assessment of Change in Wrinkles and Lines:
  Photographic Documentation: Before and after photographs will be taken to objectively compare the appearance of facial wrinkles and lines. The improvement will be graded using the following scale:
  Grade 0: No change or worsening of wrinkles. Grade 1: Slight improvement, minimal reduction in wrinkles. Grade 2: Moderate improvement, visible reduction in wrinkles. Grade 3: Significant improvement, marked reduction in wrinkles.
Facial Appearance | Upto 2 years
  Patients will provide feedback on their satisfaction with the treatment outcome and perceived changes in their facial appearance.
Assessment of Wrinkle Severity | Upto 2 years
  The WSRS will rate the severity of wrinkles on a scale of 1 to 5, with 1 indicating no wrinkles and 5 indicating severe wrinkles.

SECONDARY OUTCOMES:
Assessment of Skin Reaction | Upto 2 years
  The Principal Investigator (PI) will measure the presence and severity of skin reactions using a grading scale, where:
  Grade 0 represents no skin reaction, Grade 1 represents mild redness or inflammation, Grade 2 represents moderate redness or inflammation, and Grade 3 represents severe redness, inflammation, or swelling. By assigning a numerical value to skin reactions, the PI will quantify the degree of immune response, allowing for measurable comparisons over time.

CONTACTS AND LOCATIONS:
Overall Officials: Otis Scroggins, BS, CNA, Principal Investigator — Global Aesthetics LLC
Locations (2):
- United States (2):
  - Global Aesthetics LLC, Cisco, Texas
  - Global Aesthetics LLC, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The reason for this decision is due to ongoing considerations regarding data privacy, ethical considerations, and the need for further consultation with relevant stakeholders, including participants and regulatory bodies.